CLINICAL TRIAL: NCT00054834
Title: A Phase I Clinical Trial of Radiolabeled Immunotherapy With Humanized LL2 in Patients With Refractory or Recurrent Non-Hodgkin's Lymphoma
Brief Title: Study of 90Y-hLL2 to Treat Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL2-14
Record Dates: First submitted 2003-02-11; First posted 2003-02-13 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2008-01

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — epratuzumab

INTERVENTIONS:
Drug: hLL2 (epratuzumab)

SUMMARY:
The purpose of this trial is to determine the safety of 90Y-hLL2 at different dose levels in the treatment of Non-Hodgkin's lymphoma.

ELIGIBILITY:
Disease Characteristics:

* Patients with a documented histologic or cytologic diagnosis of B-cell NHL.
* Patients who have failed at least one regimen of chemotherapy and are not eligible for any alternate therapies of higher therapeutic priority.
* Patients with at least one measurable tumor site > 1.5 cm in at least one dimension.

Prior/Concurrent Therapy:

* Chemotherapy: Patients must have failed standard therapy or are not eligible for any alternate therapies of higher therapeutic priority.
* Biologic Therapy: Patients who have received human or humanized monoclonal antibodies will be eligible provided pre-study evaluations demonstrate no significant reactivity with hLL2 IgG (i.e., HAHA).
* Radiotherapy: No prior radiation therapy to >25% of the bone marrow. No prior radiation to maximal tolerable levels for any critical organ (e.g., 2,000 cGy for the lungs and kidneys). Patients who have had whole pelvic irradiation are not eligible.

Patient Characteristics/Inclusion Criteria:

* Age Range: Male or Female at least 18 years of age
* Performance Status: Patients with a Karnofsky performance status > 60% (or equivalent, ECOG 0-2) and expected survival of at least 12 weeks.
* Hematopoietic: Hemoglobin > 10 g/dL; ANC > 1.5x10^9/L; Platelets > 100x10^9/L;
* Hepatic: Serum bilirubin < 2.0 mg/dL; AST and ALT < 2 x ULN w/o liver metastases or <5 x ULN w/liver metastases
* Renal: Creatinine < 2.0 mg/dL
* Cardiovascular: Patients with LVEF >/= 50% by MUGA or 2D-ECHO.
* Pulmonary: Patients with DFCO and FEV1 >/= 60% by required Pulmonary Function Tests.
* Other: Patients agreeing to use a medically effective method of contraception while enrolled in the study. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the study. Patients able to understand and give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas